CLINICAL TRIAL: NCT02599597
Title: Prevention of Depressive Relapse by Means of Physical Exercise and Lifestyle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Olof Johansson, PhD student, Lund University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: rel-prev
Record Dates: First submitted 2015-11-05; First posted 2015-11-06 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Therapist-assisted iCBT (Experimental): Internet-delivered cognitive behavioral therapy (iCBT), containing physical activity and sleep management for preventing depressive relapse. Monthly depression screening with therapist feedback.
  Interventions: Behavioral: Therapist-assisted iCBT; Behavioral: Monthly screening with feedback
- Monthly screening with feedback (Active Comparator): Monthly depression screening with therapist feedback.
  Interventions: Behavioral: Monthly screening with feedback
- Control (No Intervention): No intervention, follow-up along with all participants at 6 and 12-months.

INTERVENTIONS:
Behavioral: Therapist-assisted iCBT — 13 week long individualized prevention program containing, physical activation, sleep management, tailored cognitive behavioral therapy for individual problems.
  Arms: Therapist-assisted iCBT
Behavioral: Monthly screening with feedback — Participants are screened with a depression inventory each month and receives feedback from a therapist on the results
  Arms: Monthly screening with feedback; Therapist-assisted iCBT

SUMMARY:
Depression treatments including physical activity and sleep management has been shown to relieve depressive symptoms among participants suffering depressive episodes. This study evaluates the potential of these methods as prevention of depressive relapse or recurrence

ELIGIBILITY:
Inclusion Criteria:

* A history of at least one episode of Major Depression.
* If medicating - Taking a stable (since one month) and therapeutic dosage of antidepressant medication
* Being able to read and write Swedish
* Having access to the internet

Exclusion Criteria:

* Fulfilling the criteria for Major depression
* Bipolar disorder
* Psychosis
* Substance abuse
* Suicidality
* Currently in psychotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-02; Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Depressive relapse (change in diagnostic status, SCID-I) | Baseline - 12 months
  Monthly screening via Montgomery-Asberg Depression Rating Scale - Self rated & Structured Clinical Interview for DSM IV
Change from baseline in depressive symptoms (MADRS-S) | Baseline - 6 months
  Change in depressive symptoms will be measured by an internetbased version of the Montgomery-Asberg Depression Rating Scale - Self rated.
Change from baseline in depressive symptoms (MADRS-S) | Baseline - 12 months
  Change in depressive symptoms will be measured by an internetbased version of the Montgomery-Asberg Depression Rating Scale - Self rated.
Change from baseline in depressive symptoms (MADRS-S) | Monthly, 0-12 months
  Change in depressive symptoms will be measured by an internetbased version of the Montgomery-Asberg Depression Rating Scale - Self rated.

SECONDARY OUTCOMES:
Change from baseline in health related quality of life (EQ-5D) | Baseline - 3 months
  Health related quality of life will be measured by an internet based version of the EQ-5D.
Change from baseline in health related quality of life (EQ-5D) | Baseline - 6 months
  Health related quality of life will be measured by an internet based version of the EQ-5D.
Change from baseline in health related quality of life (EQ-5D) | Baseline - 9 months
  Health related quality of life will be measured by an internet based version of the EQ-5D.
Change from baseline in health related quality of life (EQ-5D) | Baseline - 12 months
  Health related quality of life will be measured by an internet based version of the EQ-5D.
Change from baseline in Outcomes Questionnaire 45 (OQ-45) | Baseline - 3 months
  The OQ-45 measures functioning in 3 domains: Symptom distress (heavily loaded for depression and anxiety), Interpersonal functioning, and Social Role. It enables the clinician to assess functional level and change over time.
Change from baseline in Outcomes Questionnaire 45 (OQ-45) | Baseline - 6 months
  The OQ-45 measures functioning in 3 domains: Symptom distress (heavily loaded for depression and anxiety), Interpersonal functioning, and Social Role. It enables the clinician to assess functional level and change over time.
Change from baseline in Outcomes Questionnaire 45 (OQ-45) | Baseline - 9 months
  The OQ-45 measures functioning in 3 domains: Symptom distress (heavily loaded for depression and anxiety), Interpersonal functioning, and Social Role. It enables the clinician to assess functional level and change over time.
Change from baseline in Outcomes Questionnaire 45 (OQ-45) | Baseline - 12 months
  The OQ-45 measures functioning in 3 domains: Symptom distress (heavily loaded for depression and anxiety), Interpersonal functioning, and Social Role. It enables the clinician to assess functional level and change over time.
Change from baseline in the International Physical Activity Questionnaire (IPAQ) | Baseline - 3 months
  The International Physical Activity Questionnaire is a measure of physical activity
Change from baseline in the International Physical Activity Questionnaire (IPAQ) | Baseline - 6 months
  The International Physical Activity Questionnaire is a measure of physical activity
Change from baseline in the International Physical Activity Questionnaire (IPAQ) | Baseline - 9 months
  The International Physical Activity Questionnaire is a measure of physical activity
Change from baseline in the International Physical Activity Questionnaire (IPAQ) | Baseline - 12 months
  The International Physical Activity Questionnaire is a measure of physical activity
Morisky Medication Adherence Scale (MMAS-8) | Baseline - 3 months
  Self-reported measure of medication adherence
Morisky Medication Adherence Scale (MMAS-8) | Baseline - 6 months
  Self-reported measure of medication adherence
Morisky Medication Adherence Scale (MMAS-8) | Baseline - 9 months
  Self-reported measure of medication adherence
Morisky Medication Adherence Scale (MMAS-8) | Baseline - 12 months
  Self-reported measure of medication adherence
Insomnia Severity Index (ISI) | Baseline - 3 months
  Insomnia issues
Insomnia Severity Index (ISI) | Baseline - 6 months
  Insomnia issues
Insomnia Severity Index (ISI) | Baseline - 9 months
  Insomnia issues
Insomnia Severity Index (ISI) | Baseline - 12 months
  Insomnia issues
Alcohol Use Disorder Identification Test (AUDIT) | Baseline - 3 months
Alcohol Use Disorder Identification Test (AUDIT) | Baseline - 6 months
Alcohol Use Disorder Identification Test (AUDIT) | Baseline - 9 months
Alcohol Use Disorder Identification Test (AUDIT) | Baseline - 12 months
Time to depressive relapse | Baseline - 12 months
  Time to depressive relapse is recorded as secondary outcome variable
Self reported treatment seeking | Baseline - 12 months
  Treatment seeking among participants is recorded as secondary outcome variable

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Gunnar Lundh, Professor, Principal Investigator — Lund University, Departement of psychology
Locations (1):
- Vuxenpsykiatrimottagning allmänpsykiatri Fosievägen Malmö, Malmo, Skåne County, Sweden